CLINICAL TRIAL: NCT03155568
Title: Safety and Efficacy of Single Ankle, Single Popliteal or Combined Ankle and Popliteal Block for Diabetic Foot Surgery: A Comparative Study
Brief Title: Safety and Efficacy of Three Local Block Techniques for Diabetic Foot Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdel-Baky Abdel-Rahman, lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008718/ref.no2015
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia, Regional
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- sciatic nerve block (Active Comparator): ultrasound guided sciatic nerve block by injecting 30ml of 0.5% bupivacaine and visualized circumferentially spreading around the sciatic nerve
  Interventions: Procedure: sciatic nerve block; Drug: Bupivacaine
- ankle block (Active Comparator): ankle block performed by injecting 20 ml of 0.5% bupivacaine in equal amounts around the five major nerves supplying the foot
  Interventions: Procedure: ankle block; Drug: Bupivacaine
- combined popliteal and ankle block (Active Comparator): combined block performed by the use of 20 ml of 0.25% bupivacaine for sciatic nerve block followed by the ankle block with use of 20 ml of 0.5% bupivacaine both in the same manner as other two groups.
  Interventions: Procedure: sciatic nerve block; Procedure: ankle block; Drug: Bupivacaine

INTERVENTIONS:
Procedure: sciatic nerve block — sciatic nerve block at popliteal fossa
  Arms: combined popliteal and ankle block; sciatic nerve block
Procedure: ankle block — block of major nerves supplying the foot at the level of the ankle
  Arms: ankle block; combined popliteal and ankle block
Drug: Bupivacaine — blocking the lower limb nerve supply at the level of the popliteal fossa and ankle using the local anesthetic bupivacaine

SUMMARY:
Diabetic patients suffering diabetic foot disease have sever comorbidities, as hypertension, ischemic heart disease, autonomic neuropathy, infections and gastric reflux all of which contribute to a high risk profile for anesthesia.

failure rate associated with ankle or popliteal nerve block may be higher than accepted, the study hypothesized that combined ankle and popliteal block may increase the success rate with no added complications.

DETAILED DESCRIPTION:
Diabetic patients suffering diabetic foot disease regularly have sever co-morbidities, they are more liable to hypertension, ischemic heart disease, autonomic neuropathy, infections and gastric reflux all of which contribute to a high risk profile for anesthesia according to American society of anesthesiologists patients classification.

Anesthetic management for diabetic foot disease surgery is a frequent challenge and should be undertaken with a careful consideration of the anesthetic techniques available.

Hazards of general anesthesia is more likely in diabetic patients as they have low reserves to preserve against additional straining factors during general anesthesia consequently, avoiding general anesthesia in this population may be a central concern to ensure optimal peri-operative management following lower limb surgery. Neuraxial anesthesia is complicated by urinary retention, hypotension and postdural puncture headache and backache. In chronic ischemic legs, with multiple and diffuse stenosis in the leg segmental vessels, hypotension can precipitate thrombosis easily. In addition fluid loading and vasopressor administration may not be ideal methods to treat hypotension since end stage renal disease and coronary artery occlusive disease are common in these patients.

Relative to central nerve block, peripheral limb blocks are more discriminatory in their action and consequently result in less interference of bladder function and motor impairments. Also with peripheral nerve block, patients do not require postoperative fasting that help in preserving patient glycemic control. Moreover. Nerve block anesthesia has the advantages of improved postoperative pain control and it is more economical reducing hospital and associated expenses.

Ankle block alone has high failure rate and require more than usual dose to get effective. In popliteal block larger dose is needed than ankle and there is more time delay. The investigators thought to get the advantages of using local than general anesthesia with combined ankle and popliteal blocks to increase potentiation and decrease doses in diabetic foot surgery.

Aim of the study is to compare between single ankle, single popliteal and combined ankle popliteal block in diabetic patients undergoing elective foot surgery to determine block success rate, safety and efficacy to find the method of better outcome and lesser side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) II and III
* Co-operative
* Diabetic patients
* Scheduled for various types of elective diabetic unilateral foot operations

Exclusion Criteria:

* Patients suffering psychiatric neurological or neuromuscular disorders.
* Allergy to local anesthetics used.
* Infection at the block site.
* Sever renal and hepatic impairment.
* Patients receiving chronic analgesic therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-15 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
failure rate | from the time of randomization until 5 days postoperatively
  number of patients converted to general anesthesia

SECONDARY OUTCOMES:
The onset of sensory block | from the time of randomization until 5 days postoperatively
  Loss of sensation to pin- prick
The onset of motor block | from the time of randomization until 5 days postoperatively
  complete inability to move the foot
duration of sensory block | from the time of randomization until 5 days postoperatively
  duration till return in any sensation in the distribution of blocked nerve
Duration of motor blockade | from the time of randomization until 5 days postoperatively
  duration till return of motor function

CONTACTS AND LOCATIONS:
Overall Officials: Jehan S Ahmed, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided